CLINICAL TRIAL: NCT03688594
Title: Non Invasive Prenatal Test of Rare Genetic Diseases: Application to Rare Intellectual Disabilities
Acronym: DEFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6792
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Genetic Disorders in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- couple : man and pregnant women (Experimental)
  Interventions: Diagnostic Test: NIPT Test

INTERVENTIONS:
Diagnostic Test: NIPT Test — This test is based onto capture and high throw put sequencing adapted to cell free plasmatic DNA of pregnant women in order to detect point mutation present in her fetus. This approach has been previously described for others clinical applications such as liquid biopsy in cancers but not for NIPT analysis.

SUMMARY:
The aim of this study is to evaluate performances of a NIPT test based onto the study of the maternal blood to search known genetic mutations already detected in the family and potentially inherited by the fetus. This test will avoid an invasive prenatal diagnosis in those families with a known genetic risk.

The performance of this test will be evaluated in terms of sensitivity and specificity with an adapted statistic model.

Secondary objectives of the protocol are

* To adapt NIPT to small DNA quantity (5-50 ng)
* To adapt bioinformatics pipeline to low rate of mosaicism
* To develop a tool to quantify the fetal fraction
* To evaluate the robustness of the method

This test is based onto capture and high throw put sequencing adapted to cell free plasmatic DNA of pregnant women in order to detect point mutation present in her fetus. This approach has been previously described for others clinical applications such as liquid biopsy in cancers but not for NIPT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Couple (father, mother) > 18 ans
* Pregnant woman (> 12-15 weeks of gestation) with a fetal sampling needed in standard care.
* informed consent obtained
* couple affiliated to the social insurance in France

Exclusion Criteria:

* DNA extraction failure
* Absence of informed consent
* Father or mother placed under judicial protection or under guardianship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-05-22 (Estimated); Study Completion 2019-05-23 (Estimated)

PRIMARY OUTCOMES:
Detection yield of fetal paternally transmitted single nucleotid variations (SNV) in free cell maternal DNA Absence of non fetal paternally transmitted single nucleotid variations (SNV) in maternal free cell DNA (cfDNA) | Measurement will be performed at the end of the protocol (12 months)

SECONDARY OUTCOMES:
Comparison of SNV detection efficiency of several bioinformatics pipeline Robustness evaluation in function of - Fetal percent in cfDNA - Genomic region - Initial input of cfDNA | Measurement will be performed at the end of the protocol (12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France